CLINICAL TRIAL: NCT01136161
Title: Double-Blind, Randomized, Placebo-Controlled Phase II Clinical Trial to Investigate the Safety, Tolerability, and Immunogenicity of the Novel Antituberculous Vaccine RUTI® Following One Month of Isoniazid Treatment in Subjects With Latent Tuberculosis Infection
Brief Title: Clinical Trial to Investigate the Safety, Tolerability, and Immunogenicity of the Novel Antituberculous Vaccine RUTI® Following One Month of Isoniazid Treatment in Subjects With Latent Tuberculosis Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Archivel Farma S.L. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RUTISAPH2
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Latent Tuberculosis Infection; Tuberculosis
Keywords: LTBI (Latent Tuberculosis Infection); TB (Tuberculosis); Vaccine
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- RUTI 5 micrograms of FCMtb in HIV - (Experimental): n=12
  Interventions: Biological: RUTI
- RUTI 25 micrograms of FCMtb in HIV - (Experimental): n=12
  Interventions: Biological: RUTI
- RUTI 50 micrograms of FCMtb in HIV - (Experimental): n=12
  Interventions: Biological: RUTI
- RUTI Matching Placebo in HIV - (Placebo Comparator): n=12
  Interventions: Biological: RUTI Matching Placebo
- RUTI 5 micrograms of FCMtb in HIV + (Experimental): n=12
  Interventions: Biological: RUTI
- RUTI 25 micrograms of FCMtb in HIV + (Experimental): n=12
  Interventions: Biological: RUTI
- RUTI 50 micrograms of FCMtb in HIV + (Experimental): n=12
  Interventions: Biological: RUTI
- RUTI Matching Placebo in HIV + (Placebo Comparator): n=12
  Interventions: Biological: RUTI Matching Placebo

INTERVENTIONS:
Biological: RUTI — dose:5 micrograms of FCMtb (Fragmented cells of M. tuberculosis); given subcutaneously twice, on days 28 and 56.
  Arms: RUTI 5 micrograms of FCMtb in HIV +; RUTI 5 micrograms of FCMtb in HIV -
Biological: RUTI — dose:25 micrograms of FCMtb (Fragmented cells of M. tuberculosis); given subcutaneously twice, on days 28 and 56.
  Arms: RUTI 25 micrograms of FCMtb in HIV +; RUTI 25 micrograms of FCMtb in HIV -
Biological: RUTI — dose:50 micrograms of FCMtb (Fragmented cells of M. tuberculosis); given subcutaneously twice, on days 28 and 56.
  Arms: RUTI 50 micrograms of FCMtb in HIV +; RUTI 50 micrograms of FCMtb in HIV -
Biological: RUTI Matching Placebo — Placebo of the vaccine RUTI; given subcutaneously twice, on days 28 and 56.
  Arms: RUTI Matching Placebo in HIV +; RUTI Matching Placebo in HIV -

SUMMARY:
The aim of the trial is to assess the safety, tolerability and immunogenicity of two doses of RUTI® vaccine administered four weeks apart after one month pre-treatment with INH.

The trial will be double-blinded, randomized and placebo-controlled with 96 subjects (48 HIV- and 48 HIV+ subjects).

Three different RUTI® doses and placebo will be tested, randomizing assigned both in HIV+ and HIV- subjects. Each subject will be randomized to receive one of the four treatments (placebo, 5, 25, 50 μg), after completion of one month INH pre-treatment (one tablet of 300mg/day, vp.o.). Each subject will receive two administrations of the same treatment, 28 days apart. Subjects will be monitored until one month after the second inoculation with RUTI®.

DETAILED DESCRIPTION:
RUTI is a therapeutic vaccine made from virulent M.tuberculosis bacteria, grown in stressful conditions, fragmented, detoxified, heat inactivated (FCMtb) and liposomed. RUTI provides a strong humoral and cellular immune response against antigens from active growing and latent bacilli but also against structural antigens, as it has been proved in animal models of latent tuberculosis infection and in phase I clinical trial of Healthy Volunteers. The vaccine has been designed to be used against Latent Tuberculosis Infection as a therapeutic vaccine after 1-month of chemotheraputic treatment, instead the current treatment based on 6-9 months of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic adult aged 18 up to 50 years.
2. No evidence of active TB (Section 8).
3. No clinically significant finding at the discretion of the investigator.
4. Willingness to undergo an HIV test.
5. Resident in or near trial site for the duration of the trial.
6. Willingness to allow the investigators to discuss the patient's medical history with his usual doctor or HIV physician.
7. No donation of blood for 56 days prior to screening and agreement to refrain from blood donation during the trial.
8. Willing and able to provide written informed consent.
9. Positive tuberculin skin test (TST +), (≥5 mm induration) and Quantiferon TB Gold positive result (according to manufacturers instructions).
10. Reliable contraception to be used by female subjects during the clinical trial.
11. Additional inclusion criteria for HIV+ groups:

    * HIV antibody positive.
    * CD4 count ≥350 cells/mL3 on a single CD4 count at the period of screening.
    * Subjects on anti-retroviral treatment can be included if clinically stable.

Exclusion Criteria:

1. Any deviation from the normal range in biochemistry or haematology blood tests or in urine analysis that is considered to be clinically significant at the discretion of the investigator. Values of Hb, WCC, platelet count, AST/ALT and creatinine should be in a normal range accordingly to the normal laboratory values.
2. Use of any investigational or non-registered drug, vaccine, or medical device other than the trial vaccine within 30 days prior to dosing of trial vaccine, or planned use during the trial period.
3. Administration of chronic (defined as more than 14 days) immunosuppressive drugs within six months of vaccination and required throughout the duration of the trial (for corticosteroids this means prednisolone or equivalent at ≥ 0.5 mg/kg/day).
4. Female of child bearing potential who intends to become pregnant during the trial.
5. Females who are pregnant, lactating, or of child bearing potential with a blood HCG positive result 24-48 hours at the screening period, or prior to every injection of RUTI®.
6. Any AIDS defining illness according to the CDC classification system for HIV infection.
7. Presence of active (previously undiagnosed) TB or being on TB treatment.
8. Suspected or known current alcohol abuse (alcohol intake questionnaire.
9. Suspected or known substance abuse.
10. Presence of any underlying disease, specifically autoimmune disease, asthma, angioedema, bleeding disorders, uncontrolled hypertension and diabetes, and any other disease that compromises the diagnosis and evaluation of response to the vaccine, excluding HIV.
11. Administration of immunoglobulins and/or any blood products within three months prior to the planned administration of the vaccine.
12. Any history of anaphylaxis in reaction to vaccination and/or other medication.
13. Investigator assessment of lack of understanding or willingness to participate and comply with all requirements of the trial protocol.
14. Any other finding which in the opinion of the investigator would significantly increase the risk of having an adverse outcome from participating in the trial.
15. Exclusion criteria relating to INH pre-treatment

    * Weight less than 40 kg.
    * Known or suspected hypersensitivity to INH.
    * Self reported chronic liver disease or symptoms suggesting active hepatitis (jaundice, nausea, vomiting, right upper quadrant pain, dark urine, pale stools).
    * Alcohol use exceeding 28 units per week (men) or 21 units per week (women) (see alcohol intake questionnaire, Appendix 17.2).
    * History of convulsions.
    * History of psychosis.
    * Peripheral neuropathy grade 2 or greater.
    * Three months post-partum.
    * Concomitant medication with phenytoin, carbamazepine; warfarin; theophylline; disulfiram; selective serotonin re-uptake inhibitor antidepressants (e.g. citalopram, fluoxetine, paroxetine, sertraline); oral ketoconazole or itraconazole.
16. Additional exclusion criterion for HIV negative groups:

    • Any confirmed or suspected immunosuppressive or immunodeficient condition, including asplenia.
17. Additional exclusion criterion for HIV+ groups • CD4 count < 350 cells/mL3.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Local tolerability | 84 days
  The investigator will evaluate the site of injection for redness, pain, swelling, and induration and functional limitation.
  Redness, swelling and induration will be evaluated and recorded on the CRF as: 0 = absent, 1 = mild, 2 = moderate, 3 = severe. If present, the extent of the reaction will be measured in mm. Pain will be recorded, after questioning the subjects, by means of a Visual Analogue Scale (VAS from 0 to 100). The presence of abscess, ulceration or necrosis will also be evaluated, measured and adequately documented.
Focal Tolerability | 84 days
  Evaluation of the hilar lymph nodes for inflammation: An un-contrasted thoracic computerised tomographic scan will be performed to evaluate the change in size of the hilar lymph nodes.
Systemic tolerability | 84 days
  Body temperature ≥38ºC, asthenia, sweating, malaise, headache, dizziness, nausea, myalgia, arthralgia, rash and generalised pruritus
Vital Signs and physical examination | 84 days
  Blood pressure (systolic and diastolic), pulse, respiratory rate, body temperature and full physical examination will be assessed
ECG | 84 days
  The following ECG parameters will be measured: Bits Frequency Heart rate, PR, QRS, QT and QTc (Bazett) intervals. Any other anomaly on the ECG (such as U wave, ischaemia, rhythm and conduction disturbances) will be evaluated by the investigator
Laboratory Tests | 84 days
  Blood samples for serum chemistry and haematology and urine sample for urinalysis will be taken under fasting conditions for evaluation of laboratory safety parameters

SECONDARY OUTCOMES:
Immunogenicity | 63 days
  Samples to perform immunogenicity testing will be collected at specified visits. Cellular mediated immunity (ELISPOT and ELISA techniques), IFN-gama Spot Forming Units after stimulation for 18 hours with five stimuli, WHO assay (stimulating whole blood 7days with PPD) and TIGRA (TSPOT TB assay).
  Peripheral blood mononuclear cells will be frozen for future immune assays. Sera will be frozen to be further tested for the antibody-mediated immunity against M.tuberculosis antigens

CONTACTS AND LOCATIONS:
Overall Officials: André S Nell, MD, Principal Investigator — Parexel Int. Bloemfontein; Pere Joan Cardona, MD, PhD, Study Chair — Archivel Farma S.L.
Locations (3):
- South Africa (3):
  - Parexel Int. Bloemfontein, Bloemfontein
  - Parexel Int. George, George
  - Parexel Int. Port Elizabeth, Port Elizabeth

REFERENCES:
- [Background] Gil O, Diaz I, Vilaplana C, Tapia G, Diaz J, Fort M, Caceres N, Pinto S, Cayla J, Corner L, Domingo M, Cardona PJ. Granuloma encapsulation is a key factor for containing tuberculosis infection in minipigs. PLoS One. 2010 Apr 6;5(4):e10030. doi: 10.1371/journal.pone.0010030. PMID 20386605
- [Background] Cardona PJ. Revisiting the natural history of tuberculosis. The inclusion of constant reinfection, host tolerance, and damage-response frameworks leads to a better understanding of latent infection and its evolution towards active disease. Arch Immunol Ther Exp (Warsz). 2010 Feb;58(1):7-14. doi: 10.1007/s00005-009-0062-5. Epub 2010 Jan 5. PMID 20049645
- [Background] Vilaplana C, Montane E, Pinto S, Barriocanal AM, Domenech G, Torres F, Cardona PJ, Costa J. Double-blind, randomized, placebo-controlled Phase I Clinical Trial of the therapeutical antituberculous vaccine RUTI. Vaccine. 2010 Jan 22;28(4):1106-16. doi: 10.1016/j.vaccine.2009.09.134. Epub 2009 Oct 22. PMID 19853680
- [Background] Domingo M, Gil O, Serrano E, Guirado E, Nofrarias M, Grassa M, Caceres N, Perez B, Vilaplana C, Cardona PJ. Effectiveness and safety of a treatment regimen based on isoniazid plus vaccination with Mycobacterium tuberculosis cells' fragments: field-study with naturally Mycobacterium caprae-infected goats. Scand J Immunol. 2009 Jun;69(6):500-7. doi: 10.1111/j.1365-3083.2009.02251.x. PMID 19439010
- [Background] Cardona PJ. A dynamic reinfection hypothesis of latent tuberculosis infection. Infection. 2009 Apr;37(2):80-6. doi: 10.1007/s15010-008-8087-y. Epub 2009 Mar 23. PMID 19308318
- [Background] Gil O, Vilaplana C, Guirado E, Diaz J, Caceres N, Singh M, Cardona PJ. Enhanced gamma interferon responses of mouse spleen cells following immunotherapy for tuberculosis relapse. Clin Vaccine Immunol. 2008 Nov;15(11):1742-4. doi: 10.1128/CVI.00255-08. Epub 2008 Sep 30. PMID 18827194
- [Background] Guirado E, Gil O, Caceres N, Singh M, Vilaplana C, Cardona PJ. Induction of a specific strong polyantigenic cellular immune response after short-term chemotherapy controls bacillary reactivation in murine and guinea pig experimental models of tuberculosis. Clin Vaccine Immunol. 2008 Aug;15(8):1229-37. doi: 10.1128/CVI.00094-08. Epub 2008 Jun 4. PMID 18524883
- [Background] Vilaplana C, Ruiz-Manzano J, Gil O, Cuchillo F, Montane E, Singh M, Spallek R, Ausina V, Cardona PJ. The tuberculin skin test increases the responses measured by T cell interferon-gamma release assays. Scand J Immunol. 2008 Jun;67(6):610-7. doi: 10.1111/j.1365-3083.2008.02103.x. Epub 2008 Apr 4. PMID 18397200
- [Background] Cardona PJ. New insights on the nature of latent tuberculosis infection and its treatment. Inflamm Allergy Drug Targets. 2007 Mar;6(1):27-39. doi: 10.2174/187152807780077282. PMID 17352686
- [Background] Guirado E, Amat I, Gil O, Diaz J, Arcos V, Caceres N, Ausina V, Cardona PJ. Passive serum therapy with polyclonal antibodies against Mycobacterium tuberculosis protects against post-chemotherapy relapse of tuberculosis infection in SCID mice. Microbes Infect. 2006 Apr;8(5):1252-9. doi: 10.1016/j.micinf.2005.12.004. Epub 2006 Jan 27. PMID 16702016
- [Background] Cardona PJ. RUTI: a new chance to shorten the treatment of latent tuberculosis infection. Tuberculosis (Edinb). 2006 May-Jul;86(3-4):273-89. doi: 10.1016/j.tube.2006.01.024. Epub 2006 Mar 20. PMID 16545981
- [Background] Cardona PJ, Amat I, Gordillo S, Arcos V, Guirado E, Diaz J, Vilaplana C, Tapia G, Ausina V. Immunotherapy with fragmented Mycobacterium tuberculosis cells increases the effectiveness of chemotherapy against a chronical infection in a murine model of tuberculosis. Vaccine. 2005 Feb 3;23(11):1393-8. doi: 10.1016/j.vaccine.2004.09.008. PMID 15661388
- [Derived] Nell AS, D'lom E, Bouic P, Sabate M, Bosser R, Picas J, Amat M, Churchyard G, Cardona PJ. Safety, tolerability, and immunogenicity of the novel antituberculous vaccine RUTI: randomized, placebo-controlled phase II clinical trial in patients with latent tuberculosis infection. PLoS One. 2014 Feb 26;9(2):e89612. doi: 10.1371/journal.pone.0089612. eCollection 2014. PMID 24586912
- See also: Fundació Institut Investigació en Ciències de la Salut Germans Trias i Pujol homepage — http://www.germanstrias.org/
- See also: Archivel Farma, S.L. homepage — http://www.archivelfarma.com